CLINICAL TRIAL: NCT03205696
Title: A Comprehensive Community-Based Strategy to Optimize the HIV Prevention and Treatment Continuum for Youth at HIV Risk, Acutely Infected and With Established HIV Infection
Brief Title: Prevention and Treatment Continuum for Youth at HIV Risk, Acutely Infected and With Established HIV Infection
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Los Angeles LGBT Center (Other); Tulane University (Other)
Responsible Party: Principal Investigator, Karin Nielsen, Principal Investigator, University of California, Los Angeles
Other Study IDs: ATNAcuteInfection
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Anti-Retroviral Agents; Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Study site staff will store blood specimens collected in this study at least through the end of the study. In addition, as part of the informed consent process, subjects will be asked to provide written informed consent for blood specimens to be stored after the end of the study for possible future testing. The specimens of participants who do not consent to long-term storage and additional testing will be destroyed at the end of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: 36 youth with new diagnosis of acute/recent HIV as defined by laboratory assays Fiebig1-V with standard care of antiretrovirals (ARV) regimen provided by the clinician
  Interventions: Drug: Antiretrovirals
- Controls: 36 youth with newly diagnosed HIV but established HIV infection (Fiebig VI) with standard care of antiretrovirals (ARV) regimen provided by the clinician
  Interventions: Drug: Antiretrovirals

INTERVENTIONS:
Drug: Antiretrovirals — The antiretroviral (ARV) regimen provided by the clinician must follow DHHS guidelines for antiretroviral naïve adolescents and adults
  Other Names: Genvoya; Stribild

SUMMARY:
This is a strategic prospective cohort study which will measure the effects of early intensive antiretroviral therapy (ART) on the establishment and persistence of HIV-1 reservoirs and HIV-1-specific immunity in acutely /recently HIV infected youth aged 12 to 24 years as compared to newly diagnosed youth with established infection > 6 months. Participants with newly diagnosed acute /recent HIV-1 infection will be offered enrollment into the study with immediate initiation of ART which is the current standard of care.

DETAILED DESCRIPTION:
Adolescents who are displaced and living in shelters or in the streets constitute an extremely vulnerable population for acquisition of HIV infection worldwide. In the U.S., homeless youth, particularly African American Gay, Bisexual, and Transgendered Youth (GBTY), are very susceptible to substance abuse, juvenile justice contact, and acquisition of HIV and other sexually transmitted infections (STI). The displaced adolescent population is not generally amenable to routine clinic follow-up in hospital settings and potentially more easily identified through mobile outreach efforts. HIV prevalence in this group can be as high as 5.3%. While HIV incidence is unknown, high rates of concurrent exposures to other STIs, substance abuse, and survival sex suggest acute infection is likely high. Pediatric studies of HIV perinatally infected infants treated very early with potent antiretroviral therapy as well as studies of adult cohorts treated during acute infection, have shown that very early treatment of HIV is associated with control and decrease in viral reservoir burden, which is likely predictive of long term HIV control. Although early treatment has not yet been demonstrated to induce a functional cure, it has been associated with an extended period of complete viral quiescence, also known as HIV drug free remission. No studies of this kind have enrolled significant numbers of adolescents. Some studies suggest HIV reservoirs from adolescents who were recently HIV infected may be more pliable and responsive to early combined antiretroviral treatment (cART) than that of adults. Prolonged control of HIV through cART initiated following established HIV infection does not appear to impact viral reservoir size. HIV remission is not attainable in this scenario following treatment interruption, even after many years of undetectable plasma virus levels while on cART. We hypothesize that very early antiretroviral treatment of adolescents with acute HIV infection will be associated with decreased viral reservoir size, and viral reservoir size will be significantly different between adolescents with acute, recent or established HIV infection. To evaluate our hypothesis, we propose to capitalize on a current community-based strategy to initiate very prompt antiretroviral treatment many times the very day of diagnosis of HIV infection. Patients with newly diagnosed HIV infection will be offered antiretroviral treatment immediately or within a very short time by our collaborating clinical sites, and through the present study will be monitored periodically for assessment of virus load and HIV reservoir assays.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants age 12 to 24 years.
2. A positive HIV diagnostic assay following a negative HIV diagnostic assay obtained in the previous study visit (if subjects are enrolled in the high risk cohort study- Project 3) or within the last six months if not followed in Study 3. A positive HIV test at baseline for subjects who are included as part of the recently diagnosed arm. HIV diagnostic assays include POC rapid tests including 4th generation rapid assays, GeneXpert HIV qualitative assays, HIV antibody assays, and HIV RNA or DNA PCR assays.
3. Ability and willingness to provide written informed consent.
4. Willingness to initiate ART
5. Willingness of treating clinician to follow DHHS guidelines for antiretroviral naïve adolescents and adults

Exclusion Criteria:

1. Prior ART use.
2. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
3. Any acute, chronic, or recent and clinically significant medical condition that, in the opinion of the site investigator, would interfere with adherence to study requirements or jeopardize the safety or rights of the participant.
4. Chronic or recurrent use of medications that modify host immune response, e.g., oral or parenteral steroids, cancer chemotherapy.
5. Clinical treatment with an ARV regimen less effective than those recommended by DHHS HIV clinical guidelines.
6. Enrollment on a experimental ARV regimen

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Our study will be recruiting youth between the ages of 12 and 24 years with newly diagnosed HIV infection (Acute /Recent or Established HIV). The study is open to all patients within this age group with a new diagnosis of HIV infection, including pregnant women. This study will include adolescents who are displaced and living in shelters or in the streets. These homeless youth will include African American Gay, Bisexual, and Transgendered Youth (GBTY), who are very susceptible to substance abuse, juvenile justice contact, and acquisition of HIV and other sexually transmitted infections (STI).
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Amount of cell-associated HIV-1 DNA | 12 months
  To compare the amount of cell-associated HIV-1 DNA (CAHD) in 5 million blood-derived CD4+ T-cells and total PBMC (assayed by quantitative ddPCR [qPCR]) at 12 months in participants who initiated ART in Fiebig I/II versus Fiebig III/IV versus Fiebig V and those with newly diagnosed but established/chronic HIV infection with sustained suppression of plasma HIV-1 RNA.

SECONDARY OUTCOMES:
Evaluate HIV-1-specific CD4+ and CD8+ T-cells | 12 and 24 months
  To evaluate HIV-1-specific CD4+ and CD8+ T-cells by flow cytometry prior to ART initiation and while HIV-1 RNA is suppressed on ART at 12 and24 months.
Assess the amount of unspliced HIV-1 RNA | 12 and 24 months
  To assess the amount of unspliced HIV-1 RNA in 5 million blood-derived CD4+ T- cells prior to ART initiation and while HIV-1 RNA is suppressed on ART at 12, and 24 months
Assess cell-associated HIV-1 RNA to DNA ratio | 12 and 24 months
  To assess cell-associated HIV-1 RNA to DNA ratio in participants with quantifiable HIV-1 DNA prior to ART initiation and while HIV-1 RNA is suppressed on ART at 12, and 24 months
Assess the decay of HIV proviral DNA | 24 months
  To assess the decay of HIV proviral DNA by ddPCR over the observational period up to 24 months in youth with acute vs established infection.
Assess the time to undetectable HIV RNA | 24 months
  To assess the time to undetectable HIV RNA among the acute and established youth and the subsequent HIV DNA decay and HIV immune parameters over the observational period up to 24 months
Evaluate demographic and behavioral factors associated with sustained adherence to ART | 24 months
  To evaluate demographic and behavioral factors associated with sustained adherence to ART or contrarily, risk of HIV transmissibility in recently infected youth.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Nielsen, M.D., Study Chair — University of California, Los Angeles
Locations (3):
- United States (3):
  - University of California, Los Angeles, Los Angeles, California
  - Los Angeles LGBT Center, Los Angeles, California
  - Tulane University, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No